CLINICAL TRIAL: NCT02003521
Title: Impact of Lung Flute Therapy on Asthma
Status: Completed | Type: Observational
Sponsor: Medical Acoustics LLC (Industry)
Collaborators: NYSTAR (Unknown)
Responsible Party: Sponsor
Other Study IDs: 426195-4
Record Dates: First submitted 2013-11-24; First posted 2013-12-06 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: Persistent Asthma
Keywords: Lung Flute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sputum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Intervension: Lung Flute
  Interventions: Device: Lung Flute

INTERVENTIONS:
Device: Lung Flute — A low frequency wave is generated at the mouth by exhaling through a mouthpiece over a laminar surface (Reed) inside the Lung Flute®. The resulting low frequency acoustic wave that is produced travels retrograde into the lower airways and lung parenchyma and increases mucociliary clearance. Patients expel air with the force required to blow out a single candle. Patients concentrate on producing a low tone through the device while breathing in a proscribed pattern. Twenty repetitions of a single two-breath pattern are performed with the device to complete a diagnostic session.

SUMMARY:
We hypothesized that the ability of the Lung Flute to enhance mucus clearance from the lower airways could be used to improve asthma control, if the device is used on a chronic basis. The primary end point of the study is the comparison of Asthma Control Test (ACT) - a validated questionnaire for asthma control and exhaled NO before, during and after using the lung flute. Several secondary end points were assessed for efficacy and safety, including health status, spirometric lung function, "stepping down" controller therapy and daily albuterol use.

DETAILED DESCRIPTION:
This is a 3 month open label study. We plan to enroll 48 subjects with asthma at the Buffalo General Medical Center Allergy Clinic or the office of Dr. James Cumella. Inclusion criteria includes: at least 12 years of age, diagnosis of asthma and no current or previous history of smoking. Exclusion criteria includes: exacerbation of asthma or hospitalization for asthma within 8 weeks prior to enrollment, predominant chronic obstructive pulmonary disease (COPD) and bronchiectasis by clinical and/or radiological assessment, history of cough syncope, pregnant or nursing women, and inability to comply with study procedures.

ELIGIBILITY:
Inclusion Criteria:

* at least 12 years of age
* diagnosis of asthma and no current or previous history of smoking.

Exclusion Criteria:

* exacerbation of asthma or hospitalization for asthma within 8 weeks prior to enrollment
* predominant COPD and bronchiectasis by clinical and/or radiological assessment
* history of cough syncope
* pregnant or nursing women
* not fluent in English
* inability to comply with study procedures.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We are seeking patients diagnosed with asthma. All subjects will have already been screened as a consequence of their being established asthma patients at the clinical sites. Patients will be identified and screened by their attending physician who will notify the investigators. The investigators are responsible for recruiting identified subjects.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2013-11; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Impact of Lung Flute Therapy on Asthma | three months
  improvement in quality of life as measured by the validated Asthma Control Test (ACT);

SECONDARY OUTCOMES:
Impact of Lung Flute on Asthma | three months
  improvement in pulmonary functions

OTHER OUTCOMES:
Impact of Lung Flute Therapy on Asthma | three months
  * reduction in levels of exhaled nitric oxide (NO) a surrogate marker of pulmonary inflammation
  * reduction in sputum eosinophils, another surrogate marker of pulmonary

CONTACTS AND LOCATIONS:
Locations (1):
- Buffalo General Medical Center Allergy Clinic, Buffalo, New York, United States

REFERENCES:
- [Background] Fujita A, Murata K, Takamori M. Novel method for sputum induction using the Lung Flute in patients with suspected pulmonary tuberculosis. Respirology. 2009 Aug;14(6):899-902. doi: 10.1111/j.1440-1843.2009.01584.x. Epub 2009 Jul 29. PMID 19659832